CLINICAL TRIAL: NCT07295470
Title: Sleep and Activity For Eating Disorders (SAFE): a Cross-sectional and Prospective Study on the Sleep Parameters.
Brief Title: Sleep and Activity For Eating Disorders
Acronym: SAFE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09C525; 55/25 (Other: Istituto Auxologico Italiano)
Record Dates: First submitted 2025-12-01; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge Eating Disorder
Keywords: Sleep; Circadian rhythms; Eating disorders
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa; Bulimia Nervosa; Binge-Eating Disorder | interventions — Actigraphy; Blood Specimen Collection; Psychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patients with anorexia nervosa (Other): Examinations of sleep, circadian rhythms, physical activity and psychological features
  Interventions: Device: Actigraphy; Biological: Collection of biological parameters; Other: Psychological testing
- Patients with bulimia nervosa (Other): Examinations of sleep, circadian rhythms, physical activity and psychological features
  Interventions: Device: Actigraphy; Biological: Collection of biological parameters; Other: Psychological testing
- Patients with binge-eating disorder (Other): Examinations of sleep, circadian rhythms, physical activity and psychological features
  Interventions: Device: Actigraphy; Biological: Collection of biological parameters; Other: Psychological testing

INTERVENTIONS:
Device: Actigraphy — The actigraph is a non-invasive device used to measure sleep-wake rhythms based on the recording of motor activity over a 24-hour period (Acker et al., 2021). Since it is easy to handle due to its physical characteristics, it can be worn for extended periods and therefore allows the collection of data related to activity and rest phases, as well as circadian rhythms. Specifically, the use of this method allows the collection of measures relating both to daytime motor activity (i.e., intensity, duration, and circadian distribution) and to nighttime sleep (i.e., duration, sleep-onset latency, wake period, number of awakenings, efficiency index, sleep and wake times).
  Other Names: Actigraphic measurements of sleep
Biological: Collection of biological parameters — Some medical parameters will be collected, including blood pressure, heart rate, respiratory rate, blood levels of ghrelin, leptin, and orexin, as well as salivary melatonin levels.
  Other Names: Biological draws (blood and salivary)
Other: Psychological testing — Participants will be asked to complete: a) Pittsburgh Sleep Quality Index (to measure subjective sleep quality); b) Morningness-Eveningness questionnaire (to measure the chronotype); c) Body Uneasiness Test (to measure body image uneasiness); d) Body Image Task (to measure the implicit perception of body image); e) Eating Disorder Inventory-3, Binge Eating Scale, Yale Food Addiction Scale (to measure the severity of eating symptoms); f) Beck Depression Inventory - II, Hospital anxiety and Depression Scale, Social Appearance Anxiety Scale (to measure depression levels); g) State Urge to be Physically Active Questionnaire (to measure physical activity levels); h) HEXACO list of adjectives (to evaluate personality traits).
  Other Names: Psychological testing through self-report measures or instruments administered by clinicians

SUMMARY:
The SAFE (i.e., Sleep and Activity For Eating disorders) study aims to investigate the characteristics of sleep, daytime activity, and circadian rhythms in a sample of patients with eating disorders-specifically anorexia nervosa, bulimia nervosa, and binge-eating disorder-as well as the relationship between these variables and physiological parameters (i.e., body mass index, hormone levels, blood chemistry parameters) and psychological parameters (i.e., levels of depression and anxiety, body image, eating-disorder symptoms).

DETAILED DESCRIPTION:
The central aim of the study is to describe sleep characteristics in a population of patients with eating disorders (i.e., anorexia nervosa, bulimia nervosa, and binge-eating disorder) attending the Center for Eating and Nutrition Disorders of the Istituto Auxologico Italiano (Piancavallo branch) - San Giuseppe Hospital.

Sleep will be characterized through the following assessments:

1. actigraphy combined with salivary melatonin measurement;
2. collection of self-report data regarding sleep characteristics and dream content (e.g., sleep and dream diary);
3. validated self-report questionnaires assessing sleep characteristics (Pittsburgh Sleep Quality Index - PSQI) and circadian rhythms (- reduced version of the Morningness-Eveningness Questionnaire - rMEQ).

Specifically, sleep characteristics will be assessed at home, during the month preceding admission to Piancavallo (Time 0), through:

1. validated self-report questionnaires assessing sleep characteristics (PSQI) and circadian rhythms (rMEQ);
2. collection of self-report data regarding sleep characteristics and dream content (e.g., sleep and dream diary), as well as actigraphy for at least one week.

Subsequently, throughout the entire inpatient stay (Time 1: first day of admission; Time 2: midpoint of the admission - 4 weeks; Time 3: the night before discharge), patients will be monitored using actigraphy and will undergo salivary melatonin measurement on the first and last day before discharge. During the same period, daily self-report data on sleep characteristics and dream content (e.g., sleep and dream diary) will be collected.

In these same patients, in addition to age, sex, anthropometric data, and blood chemistry parameters (including ghrelin, leptin, and orexin levels), as well as ongoing pharmacological treatment, the following will be assessed: presence and severity of body image distortion (Body Uneasiness Test - BUT , and Body Image Task - BIT), mood disorders (Beck's Depression Inventory - BDI, and Hospital Anxiety and Depression Scale - HADS), social anxiety related to physical appearance (Social Appearance Anxiety Scale - SAAS), severity of the eating disorder (Eating Disorder Inventory-3 - EDI-3, Yale-Food Addiction Scale - YFAS, and Binge Eating Scale - BES), intensity of the urge to engage in physical activity (State Urge to be Physically Active Questionnaire - SUPAQ), and individual differences in the expression of personality traits (HEXACO adjectives list). Measurements obtained through these psychometric tests will be collected at three timepoints: upon admission to the unit for rehabilitation (Time 1), around the midpoint of the rehabilitation program (Time 2: 4 weeks after admission), and at discharge (Time 3).

The secondary objectives will also include the following:

* Assessing the correlation of the above parameters with the intensity, duration, and circadian distribution of daytime physical activity using actigraphy and validated scales (SUPAQ); actigraphy will also allow the evaluation of several nighttime sleep parameters: sleep duration, number of awakenings, and sleep efficiency (e.g., ratio of sleep time to time in bed);
* Assessing the relationship between sleep patterns and the degree of body image distortion as measured through the BIT, which examines body-part metrics and allows calculation of the distortion index between real body measurements and those implicitly perceived by the subject, and the BUT, an additional measure of perceived inadequacy regarding one's body;
* Assessing the influence of mood disorders measured through structured interviews and standardized questionnaires (BDI-II and HADS) on sleep characteristics and eating disorder severity in the population described above;
* Assessing the influence of chronotype (e.g., morning, evening, or intermediate), investigated through the rMEQ questionnaire, on eating disorder symptomatology and on the expression of different personality traits, assessed through self-report questionnaires (HEXACO).

ELIGIBILITY:
Inclusion Criteria:

* a) Age over 18 and under 65;
* b) Diagnosis of anorexia nervosa, bulimia nervosa, or binge-eating disorder, as indicated by DSM-5-TR criteria;
* c) Adherence to the rehabilitation program.

Exclusion Criteria:

* a) Presence of severe bradycardia (BPM < 35);
* b) Severe malnutrition (BMI < 10);
* c) Presence of severe psychopathology other than the eating disorder (e.g., schizophrenia);
* d) Need to modify psychotropic or sleep-inducing pharmacological therapy during the rehabilitation program.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency (SE) | A week before the rehabilitation recovery (Time 0), at the beginning of the recovery (Time 1), half of the recovery (Time 2 - after 4 weeks from Time 1) and at the end of the recovery (Time 3 - 7 weeks from Time 1).
  Sleep efficiency will be detected through actigraphic measurements and will be compared either within and among groups.
Chronotype | A week before the rehabilitation recovery (Time 0), at the beginning of the recovery (Time 1), half of the recovery (Time 2 - after 4 weeks from Time 1) and at the end of the recovery (Time 3 - 7 weeks from Time 1).
  Chronotype is the propensity for the individual to engage in certain activities (i.e., sleep) at a particular time during a 24-hour period. It will be detected through a self-report measure, the Morningness-Eveningness Questionnaire, in its reduced version. The scale is composed by 5 items evaluating: a) preferred time for waking up, b) preferred time for going to bed, c) subjective peak alertness during the day, d) ease of getting out of bed, and e) self-assessment of being a "morning" or "evening" type. The total score ranges from 4 to 26, with the following threshold and interpretation: a) 4-10: Evening type, b) 11-18: Intermediate type, c) 19-26: Morning type.
Orexin Levels | At the beginning of the recovery (Time 1) and at the end of the recovery (Time 3 - 7 weeks from Time 1).
  Levels of orexin detected through blood exams.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi De Gennaro, Study Director — University of Roma La Sapienza; Leonardo Mendolicchio, MD, Study Director — Istituto Auxologico Italiano; Serena Scarpelli, PhD, Study Director — University of Roma La Sapienza
Locations (1):
- Istituto Auxologico Italiano - S. Giuseppe Hospital, Verbania, VB, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP